CLINICAL TRIAL: NCT05735171
Title: Tailored Supramarginal Resection in Glioblastoma Guided by Artificial Intelligence-based Recurrence Probability Maps. A Non-randomized Pilot Study
Brief Title: Supramarginal Resection in Glioblastoma Guided by Artificial Intelligence
Acronym: SupraGlio-AI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital del Rio Hortega (Other)
Collaborators: UiT The Arctic University of Norway (Other); University Hospital of North Norway (Other); University of Valladolid (Other)
Responsible Party: Principal Investigator, Santiago Cepeda, Principal Investigator, Hospital del Rio Hortega
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-PI208
Record Dates: First submitted 2023-02-07; First posted 2023-02-21 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AI-guided resection (Experimental): Tailored supramarginal surgery guided by AI-based recurrence probability maps. Aim of supramarginal resection, where the high-risk of recurrence areas identified by the AI-based model are subsidiary to be removed as safe locations for the patient.
  Interventions: Procedure: AI-guided surgery

INTERVENTIONS:
Procedure: AI-guided surgery — Neuronavigated targeted biopsy sampling. Supramarginal resection including high-risk areas of recurrence defined by a radiomics-based model.

SUMMARY:
Glioblastomas are the most common and poorly prognostic primary brain neoplasms. Despite advances in surgical techniques and chemotherapy, the median survival time for these patients remains less than 15 months. This highlights the need for more effective treatments and improved prognostic tools. The globally accepted surgical strategy currently consists of achieving the maximum safe resection of the enhancing tumor volume. However, the non-enhancing peritumoral region contains viable cells that cause the inevitable recurrence that these patients face. Clinicians currently lack an imaging tool or modality to differentiate neoplastic infiltration in the peritumoral region from vasogenic edema. In addition, it is not always feasible to include all the T2-FLAIR signal alterations surrounding the enhancing tumor in the surgical planning due to the proximity of eloquent areas and the higher risk of postoperative deficits.

However, the investigators have developed a model to predict regions of recurrence based on machine learning and MRI radiomic features that have been trained and evaluated in a multi-institutional cohort.

The investigators aim to analyze whether an adjusted supramarginal resection guided by these new recurrence probability maps improves survival in selected patients with glioblastoma.

DETAILED DESCRIPTION:
The SupraGlio-AI study aims to test the feasibility of the proposed AI-guided tailored supratotal resection for glioblastomas. The study will provide preliminary data on the accuracy of the AI model in predicting recurrence and the impact of using this information in surgical planning. This information will be crucial in determining the potential for a larger, randomized controlled trial in the future. The pilot study will also allow for refinement of the study design, intervention, and data collection processes before a larger-scale study is conducted. In addition to testing the feasibility and efficacy of the AI-guided tailored supratotal resection, this pilot study also has two secondary objectives: 1) Survival Analysis: The survival analysis will provide insights into the impact of using the AI model on patient outcomes and help determine the potential benefits of this approach. 2) Histopathological and Transcriptomic Analysis: The study will also include a histopathological and transcriptomic analysis of the tissue samples obtained from the high-risk regions defined by the AI model. This analysis will provide information on the molecular and cellular changes occurring in these regions and may offer insights into the underlying biology of glioblastoma recurrence. These data will inform the development of future studies aimed at improving patient outcomes.

By incorporating these secondary objectives, this pilot study will contribute to a more comprehensive understanding of the potential benefits of using AI in guiding tailored supratotal resection for glioblastomas. The results will inform future research and potentially lead to the development of improved treatment approaches for patients with this type of brain tumor.

ELIGIBILITY:
Inclusion Criteria:

* A suspected diagnosis of supratentorial glioblastoma by MRI.
* Tumor in non eloquent brain region according to the UCSF (University of California, San Francisco) classification, including the sensor motor areas (precentral and postcentral gyri), perisylvian language areas in the dominant hemisphere (superior temporal, inferior frontal, and inferior parietal gyri), basal ganglia, internal capsule, thalamus, and visual cortex around the calcarine sulcus
* Indication for surgical treatment and where supramarginal resection is considered possible according to the preoperative imaging. This consideration needs to be verified by two specialists in neurosurgery. This criterion needs to be verified by two senior neurosurgeons.
* Karnofsky Performance Score ≥ 70;
* Written informed consent

Exclusion Criteria:

* Tumors in eloquent areas.
* Recurrent gliomas (except biopsy)
* MR image data not usable due to artifacts during acquisition. Inability to give written informed consent
* KPS < 70
* Severe comorbidity.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Feasibility using eligibility | Screening/Enrollment
  Among all screened patients, the proportion of patients who meet the eligibility criteria
Feasibility using the proportion of consent | Screening/Enrollment
  Among all screened patients, the proportion of patients consenting to participate

SECONDARY OUTCOMES:
Efficacy using overall survival | From date of surgery until the date of death from any cause, assessed up to 36 months
  Measured in days from surgery to the time of death
Efficacy using progression-free survival | From date of surgery until the date of first documented progression, assessed up to 36 months
  Assessment of progression-free survival based on the Modified Criteria for Radiographic Response Assessment in Glioblastoma (mRANO) criteria.
Safety using the neurological function | 30 days
  The National Institutes of Healt Stroke Scale (NIHSS) will be used to assess neurological function. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment.
Safety using global disability | 30 days
  The modified Rankin scale (mRS ) is a measure of global disability that has been widely used to assess outcome after stroke. The scale runs from 0-6, running from perfect health without symptoms to death
Extent of resection | < 72 hours after surgery
  Volumetric measurement of contrast enhancement and T2-FLAIR signal alteration on MRI
Postoperative complication | 30 days
  Relevant post surgical complication that requires a second surgery or prolong the length of hospitalization (i.e. hematoma, infection)

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Cepeda, PhD, Principal Investigator — Hospital Río Hortega
Locations (1):
- University Hospital Rio Hortega, Valladolid, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cepeda S, Luppino LT, Perez-Nunez A, Solheim O, Garcia-Garcia S, Velasco-Casares M, Karlberg A, Eikenes L, Sarabia R, Arrese I, Zamora T, Gonzalez P, Jimenez-Roldan L, Kuttner S. Predicting Regions of Local Recurrence in Glioblastomas Using Voxel-Based Radiomic Features of Multiparametric Postoperative MRI. Cancers (Basel). 2023 Mar 22;15(6):1894. doi: 10.3390/cancers15061894. PMID 36980783